CLINICAL TRIAL: NCT00942019
Title: Bronchial Inflammation in Adolescent Smokers With and Without Obesity
Brief Title: Study of Bronchial Inflammation in Adolescent Smokers With and Without Obesity
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Stefan Zielen, Goethe-University, Frankfurt, Germany
Other Study IDs: KGU-88/08
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Obesity; Tobacco Smoking
Keywords: BMI; obesity; CO; tobacco smoking; adolescents
MeSH Terms: conditions — Obesity; Tobacco Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum: total IgE, RAST urin: cotinine, leukotrienes sputum: leukotrienes, white cells whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- obese smokers: BMI > 30 kg/m2 CO ≥ 15 ppm
- non-obese smokers: BMI < 25 kg/m2 CO ≥ 15 ppm
- obese non-smokers: BMI > 30 kg/m2 CO ≤ 6 ppm
- non-obese non-smokers: BMI < 25 kg/m2 CO ≤ 6 ppm

SUMMARY:
The investigators want to assess differences in lung function and bronchial inflammation of young smokers and non-smokers with (BMI > 30) and without obesity (BMI < 25)(4 patient groups). The aim of the study is to compare differences in lung function (VC, FEV1, VC/FEV1, metacholine challenge) and bronchial inflammation in relation with smoking history and levels of exhaled CO. For the latter the investigators will analyze the levels of IL-8, IL-6, TNF alpha and INF gamma and mRNA of LBP, TLR2 and TLR4 in sputum. Further, inflammatory markers e.g. low CRP and inflammatory cytokines levels in the blood will be investigated. The aim is to describe a early stage of chronic obstructive pulmonary disease caused by cigarette smoke in juvenile smokers, and the relationship between bronchial inflammation and obesity in adolescents.

DETAILED DESCRIPTION:
Tobacco smoke is the crucial factor at the beginning and in the course of the bronchial inflammation leading to COPD. It has been shown that cigarette smoke in vitro leads to a MAP kinase and NF-κB-dependent increase of pro-inflammatory cytokines, and inhibits bacteria-induced expression of β-defensins. Several studies revealed an increase of inflammatory cytokines like IL-8 and TNF in the sputum of smokers. Further studies demonstrated an up regulation of LTB4 and LBP possibly due to the LPS derived from tobacco smoke. Hasday et al could show that up to 15 ng per cigarette LPS is released. In principle, the cigarette smoke exposure liked a mild LPS inhalation. In separate work, we could show that LPS inhalation in healthy non-smokers to an increase of CRP and LBP concentrations in the serum lead. In another study of adolescents, 24 smokers (age 17.7 years) and 24 non-smoking (age 17.5 years) were compared. The CO in smokers was significantly increased, and the NO concentrations decreased. At the same time there was a significantly greater bronchial hyperreagibility in the smoker group.

According to a recent study in Germany (KiGGS study), already 31% of the adolescents' boys and 32% of the girls do smoke. The social status is of great importance. Boys and girls from families with a low social status smoke more frequently than those from families with middle-and especially with higher social status. Similarly obesity is linked to the social status with overweight occurring more often in families with a lower social status.

A visceral obesity is closely associated with the risk of type-2-diabetes as well as other aspects of the metabolic syndrome. However, the existing insulin resistance is of fundamental importance. Due to increased visceral fat depots and subsequently increased release of proinflammatory proteins various complications do occur.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age between 14 and 22 years
* smokers CO ≥ 15 ppm
* non-smokers CO ≤ 6 ppm

Exclusion Criteria:

* Asthma > GINA I°
* others chronic diseases or infections (e.x. HIV, tuberculosis, malignancy)
* pregnancy
* therapy with systemic corticosteroids
* permanent treatment with inhaled corticosteroids
* documented alcohol, substance, and/or drug abuse
* incapability to perform all study procedure

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Youth
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Bronchial inflammatory in adolescents smokers with and without obesity | one day

SECONDARY OUTCOMES:
Association of bronchial inflammatory parameters in sputum and in the blood | one day

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof., Principal Investigator — Children´s Hospital, Goethe-University, Frankfurt, Germany
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt am Main, Germany

REFERENCES:
- [Background] Karimi K, Sarir H, Mortaz E, Smit JJ, Hosseini H, De Kimpe SJ, Nijkamp FP, Folkerts G. Toll-like receptor-4 mediates cigarette smoke-induced cytokine production by human macrophages. Respir Res. 2006 Apr 19;7(1):66. doi: 10.1186/1465-9921-7-66. PMID 16620395
- [Background] Carpagnano GE, Kharitonov SA, Foschino-Barbaro MP, Resta O, Gramiccioni E, Barnes PJ. Increased inflammatory markers in the exhaled breath condensate of cigarette smokers. Eur Respir J. 2003 Apr;21(4):589-93. doi: 10.1183/09031936.03.00022203. PMID 12762340
- [Background] Garey KW, Neuhauser MM, Robbins RA, Danziger LH, Rubinstein I. Markers of inflammation in exhaled breath condensate of young healthy smokers. Chest. 2004 Jan;125(1):22-6. doi: 10.1378/chest.125.1.22. PMID 14718416
- [Background] Csoma Z, Kharitonov SA, Balint B, Bush A, Wilson NM, Barnes PJ. Increased leukotrienes in exhaled breath condensate in childhood asthma. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1345-9. doi: 10.1164/rccm.200203-233OC. Epub 2002 Sep 5. PMID 12406853
- [Background] Sebastian A, Pehrson C, Larsson L. Elevated concentrations of endotoxin in indoor air due to cigarette smoking. J Environ Monit. 2006 May;8(5):519-22. doi: 10.1039/b600706f. Epub 2006 Mar 27. PMID 16688352
- [Background] Kitz R, Rose MA, Borgmann A, Schubert R, Zielen S. Systemic and bronchial inflammation following LPS inhalation in asthmatic and healthy subjects. J Endotoxin Res. 2006;12(6):367-74. doi: 10.1179/096805106X153934. PMID 17254391
- [Background] KiGGS Study of Robert Koch Institut
- [Background] Kornmann O et al. Influence of second hand tobacco smoke exposure on inflammatory parameters in induced sputum Abstract ATS 2008